CLINICAL TRIAL: NCT04276220
Title: Prevalence of Wild-Type Transthyretin Cardiac Amyloidosis Among Patients Undergoing Carpal Tunnel Release Surgery - A Prospective Study
Brief Title: Prevalence of wtATTR-CM After Carpal Tunnel Release Surgery
Acronym: CACTuS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, DMSc, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-178-19
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Transthyretin Amyloidosis; Transthyretin Cardiac Amyloidosis; Wild-Type Transthyretin-Related (ATTR)Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tenosynovial Biopsy (Other)
  Interventions: Diagnostic Test: Tenosynovial biopsy

INTERVENTIONS:
Diagnostic Test: Tenosynovial biopsy — Tenosynovial biopsy taken from the wrist at the carpal tunnel release surgery.

SUMMARY:
Patients above the age of 60 will be recruited at their carpal tunnel release surgery. Biopsies will be taken from the wrist and examined for the presence of amyloid protein. A amyloid-positive biopsy will refer the patients for cardiac examination including blod- and urine samples examined for transthyretin.

If the result of the cardiac examination is suspected cardiac amyloidosis, the patient will be referred for a diagnostic TC99-DPD scintigraphy. If the scintigraphy is positive, the patient will be referred for right heart catherization (RHC) and an exercise test.

Myocardial biopsies will be taken at the RHC and examined with electron microscopy and high resolution respirometry.

ELIGIBILITY:
Inclusion Criteria:

* Males above 65 years of age, females above 75 years of age.
* Scheduled idiopathic carpal tunnel release surgery.
* Informed written consent.

Exclusion Criteria:

* Operation by other indication, e.g.
* Fracture
* Ganglion
* Known amyloidosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of wild-type transthyretin cardiac amyloidosis in patients undergoing surgery for idiopathic Carpal Tunnel Syndrome Surgery where biopsies from transverse carpal ligament stain positive for amyloid. | Through study completion, 6 years.
  We will examine the amyloid deposits prevalence in biopsies from the Carpal Tunnel and ATTRwt prevalence in an aged and predominantly male population operated for idiopathic Carpal Tunnel Syndrom. Diagnosis of wild-type cardiac amyloidosis will be determined by TC99-DPD scintigraphy, endomyocardial biopsy, or both. Biopsies will be examined using Congo Red staining and fluorescent light

SECONDARY OUTCOMES:
Levels of transthyretin in blood and urine from patients with suspected wild-type transthyretin cardiac amyloidosis | Has been added after study start, will run through study completion, 3 years.
  We will investigate the plasma and urine levels of different forms of TTR (total TTR, misTTR, and fragTTR) in patients with amyloid deposits in the transverse carpal ligament, patients subsequently diagnosed with ATTRwt-CM and in patients with already diagnosed ATTRwt matched age and gender.
  We will investigate whether the levels of TTR is higher among ligament amyloid positive patients that are subsequently diagnosed ATTRwt-CM as compared to those without ATTR-CM.
Comparing patients diagnosed with wild-type transthyretin cardiac amyloidosis due to screening with age and gender matched clinically diagnosed ATTRwt patients. | Through study completion, 6 years.
  Compare NAC-stage, NYHA-class, LVEF ect.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No